CLINICAL TRIAL: NCT01864967
Title: Carbon Dioxide Infusion:Clinical and Histological Appraisal in Chronic Wounds
Status: Completed | Type: Observational
Sponsor: Institute of Assistance in Plastic Surgery, Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: AC-001
Record Dates: First submitted 2008-11-23; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-01

CONDITIONS: Wounds
Keywords: carbon dioxide infusion; dilatation of peripheral blood vessels; capillaries; macrophags; fibroblasts; Improvement granulation tissue in chronic wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- carbon dioxide infusion: Group I: receive carbon dioxide infusion
- control: did not receive carbon dioxide

SUMMARY:
Carbon dioxide infusion is a non surgical procedure applied via percutaneous, transdermal and subcutaneous. Increase in the concentration of carbon dioxide decreases pH activating local nitric oxide that stimulates collateral vessels formation, vascular endothelial growth factor and basic fibroblast growth factor. Carbon dioxide infusion restores the blood flow in chronic wounds of the lower limbs.

DETAILED DESCRIPTION:
Ten patients with chronic wounds caused by venous insufficiency at both lower limbs were distributed into groups. Group I was composed by wounds in the right lower limb that received carbon dioxide and group II by wounds in the left lower limb that not received carbon dioxide, both related to the same patient. Carbon dioxide infusion was performed with the needle pointed toward the granulation tissue, 5cm distant from each one at intervals of 4 days. Biopsies were collected from the wounds before carbon dioxide infusion and after the 3rd, 5th and 10th application. Statistical analysis of the data was performed using Wilcoxon's test and Friedman's variance analysis and multiple comparisons test.

ELIGIBILITY:
Inclusion Criteria:

* chronic wounds caused by venous insufficiency

Exclusion Criteria:

* other diseases of the lower limbs

Ages: 49 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 10 patients with chronic wounds on both lower limbs
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
dilatation of peripheral blood vessels, number of capillaries, macrophages and fibroblasts | 10 sessions (5 weeks) per patient

CONTACTS AND LOCATIONS:
Overall Officials: Antonio CA Abramo, PhD M.D., Study Chair — ACA Institute of Assistance in Plastic Surgery Sao Paulo
Locations (1):
- Instute of Assistance in Plastic Surgery of São Paulo, São Paulo, São Paulo, Brazil